CLINICAL TRIAL: NCT05198700
Title: The Effect of a Probiotic on Symptoms of Infantile Colic: a Randomized, Double-blind, Placebo-controlled Study (PROCOLIN)
Brief Title: The Effect of Probiotics on Symptoms of Infantile Colic
Acronym: PROCOLIN
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Null recruitment
Sponsor: Lallemand Health Solutions (Industry)
Collaborators: ProbiSearch SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: L-022
Record Dates: First submitted 2021-12-03; First posted 2022-01-20 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-02

CONDITIONS: Colic
Keywords: Infantile colic; Crying time; Probiotics; Sleep duration
MeSH Terms: conditions — Colic

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants in this group will be randomized to receive the probiotic formulation for 4 weeks.
  Interventions: Dietary Supplement: Probiotic Formulation
- Control Group (Placebo Comparator): Participants in this group will be randomized to receive the placebo for 4 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic Formulation — Participants will be asked to take one sachet daily, containing 1 billion CFU of the probiotic formula. Sachets must be dissolved in warm water or mother's milk before consumption.
  Arms: Experimental Group
Dietary Supplement: Placebo — Participants will be asked to take one sachet containing the placebo daily. Sachets must be dissolved in warm water or mother's milk before consumption.
  Arms: Control Group

SUMMARY:
The aim of this study is to evaluate the effects of a probiotic formulation on the daily crying patterns of infants. It is hypothesized that participants given the probiotic formulation will show a significant reduction in daily crying duration compared to participants receiving the placebo.

DETAILED DESCRIPTION:
Participants diagnosed with symptoms of infantile colic will be recruited to participate in this randomized, double-blind, placebo-controlled, two-arm parallel study. Eligible participants will be enrolled in this study for 6 weeks, and will undergo a 1-week run-in baseline period followed by a 4-week interventional period, then a 1-week follow-up period.

The study will consist of 7 visits (V0 to V6): 4 in-person visits that alternate with 3 phone calls.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female.
2. Age ≤ 8 weeks old.
3. Diagnosis of infantile colic according to the Rome IV criteria. Infants must show cry or fuss behaviour for 3 or more hours per day, during 3 or more days in 7 days.
4. Exclusively breastfeeding and planning to breastfeed for duration of study.
5. With a written informed consent signed by the father, mother, or legal guardian, and with expressed or implied consent of the other parent.
6. With parents willing to complete questionnaires, records, and diaries associated to the study and to complete all clinical visits and telephone calls.

Exclusion Criteria:

1. Birthweight < 2500 g.
2. Gestational age < 37 weeks.
3. Apgar score at 5 minutes < 7.
4. Partially or fully formula fed infants, with the exception of the first 4 days after birth.
5. Stunted growth/weight loss (< 100 g/week from birth to last reported).
6. Gastroesophageal reflux disease, short bowel syndrome, chronic intestinal diseases or gastrointestinal malformations.
7. Fever and/or infectious diseases, or current systemic infections, or history of congenital infections.
8. Genetic diseases and chromosomal abnormalities.
9. Metabolic diseases or pancreatic insufficiency.
10. Immunodeficiency.
11. Neurological diseases.
12. Suspected or confirmed food allergies and intolerances.
13. Use of probiotics, prebiotics, antibiotics, or gastric acid inhibitors by the infant at any time from birth to the moment of screening.
14. Use of anti-colic medication at any time from birth to the moment of screening.
15. Use of probiotic supplements by the mother between the birth of their infant and the moment of screening.
16. Currently enrolled in another clinical study or having participated in another clinical trial from birth to the moment of screening.

Max Age: 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Symptoms of infantile colic | 5 weeks
  Comparison of the difference in the proportion of infants with reductions in mean daily crying duration by over 50 percent from baseline between the probiotic and placebo groups, as assessed by the baby's Daily Diary.

SECONDARY OUTCOMES:
Symptoms of infantile colic: Daily crying duration | 5 weeks
  Comparison of the average change from baseline in the mean daily crying duration between the probiotic and placebo groups, as assessed by the baby's Daily Diary.
Symptoms of infantile colic: Number of crying episodes | 5 weeks
  Comparison of the change in the number of crying episodes from baseline between the probiotic and placebo groups, as assessed by the baby's Daily Diary.
Symptoms of infantile colic: Sleep duration | 5 weeks
  Comparison of the difference in sleep duration from baseline between the probiotic and placebo groups, as assessed by the baby's Daily Diary.
Symptoms of infantile colic: Time to a 25 and 50 percent reduction in cry/fuss time | 5 weeks
  Comparison of the difference in time to reach a 25 percent and 50 percent improvement in cry/fuss time from baseline between the probiotic and placebo groups, as assessed by the baby's Daily Diary.
Symptoms of infantile colic: Parental perception | 5 weeks
  Comparison of the difference in the perceived evolution of colic symptoms by parents of participants in the probiotic and placebo groups, as assessed by questions about the evolution of colic symptoms at visits 2 and 4.
Change in the mother's quality of life | 5 weeks
  Comparison of the changes in the overall score of the SF-36 from baseline (0 to 100; a higher score corresponds to a better quality of life), between mothers of participants in the probiotic and placebo groups.
Bowel movement frequency | 5 weeks
  Comparison of the changes in bowel movement frequency and consistency from baseline between the probiotic and placebo groups, as assessed by the Amsterdam Infant Stool Scale.
Fecal strain recovery of the probiotic | 5 weeks
  Presence of the probiotic strain in participants in the probiotic group, as determined by qPCR analysis of stool samples collected at baseline and at week 4.
Fecal microbiome composition | 5 weeks
  Comparison of the differences in the composition of fecal microbiota and mycobiota between the probiotic and placebo groups, as determined by 16S sequencing of stool samples collected at baseline and at week 4.

OTHER OUTCOMES:
Fecal protein markers | 5 weeks
  Comparison of the differences in the concentration of fecal protein markers between probiotic and placebo groups in stool samples collected at baseline and at week 4. Proteins will be quantified using immunoassay methods.
Incidence of Adverse Events | 6 weeks
  Comparison of the number of adverse events (AEs) and serious adverse events (SAEs) recorded in the probiotic and placebo groups.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Jiménez Quintana, Ph.D., Study Director — ProbiSearch SL
Locations (5):
- Spain (5):
  - Centro de Salud Cerro del Aire, Majadahonda, Madrid
  - Centro de Salud Ibiza, Madrid
  - Hospital Vithas La Milagrosa, Madrid
  - Centro de Salud Campo de la Paloma, Madrid
  - Hospital Vithas Aravaca, Madrid

IPD SHARING:
Plan to Share IPD: No
After publications of the results, de-identified data will be shared with qualified researchers and scientists upon reasonable request to the sponsor including a detailed proposal of the intended use of the data, as per the Lallemand Health Solutions Inc. Policy on Clinical Trial Transparency and Data Sharing (available upon request).